CLINICAL TRIAL: NCT06179771
Title: HA380 Column Use in Critically Ill Patients Receiving Extracorporeal Support for Acute Critical Illness; a Prospective, Randomised, Interventional, Feasibility, Pilot Study (HACEC)
Brief Title: Pilot Study on HA380 Column Use in Critically Ill Patients Receiving Extracorporeal Support.
Acronym: HACEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Jafron Biomedical Company Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160716; 340810 (Other: IRAS)
Record Dates: First submitted 2023-10-09; First posted 2023-12-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-12

CONDITIONS: Acute Kidney Injury; ARDS; Inflammation; Extracorporeal Circulation; Complications
MeSH Terms: conditions — Acute Kidney Injury; Inflammation

STUDY DESIGN:
Intervention Model Description: Consecutive study participants would be assigned using block randomisation into the intervention arm or the standard of care arm. Patients in the intervention arm would be treated with the HA380 column. The outcomes would be compared with patients who received standard ICU care .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Active Comparator): Patients assigned to interventional arm will receive treatment with a cytokine adsorption device (HA 380) within 72 hours of being admitted to ICU. This is in addition to standard evidence based ICU care. Each patient will receive 2 treatments each lasting a maximum of 6 hours in a 24 hour period.
  Interventions: Device: HA 380
- Standard care (No Intervention): Patients assigned to the standard care arm would receive evidence based standard ICU care.

INTERVENTIONS:
Device: HA 380 — HA380 hemoperfusion cartridge is filled with neutral macroporous resin, mainly adsorbing molecules from 10 to 60 kDa. Because of the accurate 3D macroporous structure and over 54000 m2 adsorption surface area of the resin. The cartridge is attached to the extracorporeal circuit in series with the oxygenator/ filter of the extracorporeal circuit.
  Arms: Interventional

SUMMARY:
Patients who are very ill either due to a severe infection, major organ injury, trauma or a major operation may require significant support with devices such as a dialysis machine for the kidneys or Extracorporeal Membrane Oxygenation (ECMO) for the heart and lungs. This is often due to a reaction of the body to the insult which is termed inflammation. The investigators would like to assess if the use of a device that can remove the agents driving this reaction can lead to a quicker recovery form the illness. The device is a blood filter called HA380 and it would be connected to either the dialysis machine or the ECMO circuit. The investigators want to assess the feasibility of conducting a study with the HA380 column. We will also evaluate if the use of the HA380 column has an effect on the time spent on dialysis or ECMO, time spent on the breathing machine, time spent requiring drugs to support blood pressure and time spent in the intensive care unit.

DETAILED DESCRIPTION:
The role of inflammation in the pathophysiology of major organ dysfunction in critically ill patients is well established and this correlates with the degree of organ dysfunction which consequently may require increased level of organ support in the intensive care unit. Critically ill patients present in a spectrum of inflammatory states and on the extreme end of this spectrum are patients requiring renal replacement therapy and ECMO support. This subgroup of critically ill patients have been found to have high mortality.

The concept of attenuating severe hyperinflammatory response is sometimes used in certain disease states using agents such as intravenous corticosteroids, plasma exchange and more recently, anti-cytokine monoclonal antibodies. However, these strategies are associated with side effects (e.g. Bleeding and increased risk of infection), and are not necessarily appropriate in all critically ill patients with severe inflammation. Studies investigating the efficacy of these strategies have failed to show any clinical benefit except in the setting of COVID 19 infection.1-4 Early use of cytokine adsorption devices may provide an alternative non- pharmacological pathway with fewer side effects which can be deployed early.

The most studied cytokine adsorption device is the CytoSorb column which consists of biocompatible polymer sorbent beads. Several studies have demonstrated a reduction in vasopressor requirements, IL-6 levels, and Sequential Organ Failure Assessment (SOFA) scores.5,6 However, this observation did not translate into outcome benefit. There is considerable heterogeneity in how the cytokine adsorption is delivered in these studies and the study designs. An international registry analysis did not demonstrate a mortality benefit with CytoSorb either.7

The HA380 column consists of styrene divinylbenzene copolymers. In a recent study consisting of patients undergoing cardio-pulmonary bypass, patients who received the HA 380 column required lower vasopressor doses, shorter duration of invasive mechanical ventilation and had a shorter ICU length of stay.8 A direct in- vitro comparison of the CytoSorb device and the HA 380 device shows that the latter is less efficient at removing cytokines compared to the CytoSorb device but both devices were efficient at removing pro-inflammatory cytokines.9 The role of cytokines in critical illness is a double-edged sword10, and this may well be where CytoSorb may have a disadvantage - providing higher cytokine clearance for a longer period.

We hypothesise that the HA380 column use in critically ill patients with inflammation receiving renal replacement therapy or ECMO is associated with an improvement in mortality. It is recommended to be used early (within 72 hours of commencement of extracorporeal support). HA380 hemoperfusion cartridge, mainly adsorbs molecules from 10 to 60 kDa. Because of the accurate 3D macroporous structure and over 54000 m2 adsorption surface area of the resin.HA380 haemoperfusion therapy can provide a new regimen in controlling inflammatory cytokines storm. Studies have demonstrated the ability of the HA380 column to reduce the concentration of pro-inflammatory cytokines IL-1, TNF-alpha. 11,12

The aim of this feasibility pilot is to assess the feasibility of the early use of the HA380 cytokine adsorption column in a study and its effect on the time-to-liberation from extracorporeal membrane oxygenation (ECMO) support, vasoactive drug requirement and duration of vasoactive therapy, and mortality (or clinical surrogates for all-cause mortality).

ELIGIBILITY:
Inclusion Criteria

* Consent obtained
* Male or Female, aged 18 years - 65 years.
* Admitted with a diagnosis of sepsis (according to sepsis-3 definition), trauma, ARDS of infectious or non-infectious aetiology, trauma or after major surgery
* Need for extracorporeal support and specifically renal replacement therapy (RRT) and/or ECMO.
* Vasopressor or inotropic therapy requirement at the time of RRT or ECMO support
* Within 72 hours of requiring extracorporeal support
* At least one of:
* CRP > 100 mg/L (in the absence of immunosuppressive therapy/immunomodulation)
* Lactate >2 mmol/L

Exclusion Criteria

* The participant may not enter the trial if ANY of the following apply:
* Unable to obtain consent.
* Expected to die in the next 24 hours.
* Pre-existing chronic kidney disease - requiring dialysis /eGFR < 30ml/min/1.73m2
* Pre-existing severe respiratory failure - e.g., requiring home oxygen/ home nebulisers/ poor exercise tolerance
* Chronic heart failure - NYHA class III and above
* Pregnancy
* Requirement for immediate immune modulation e.g., plasma exchange, high dose steroids , IV immunoglobulins (does not include vasoplegic dose of steroids or immune modulation for COVID 19)
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Successful use of HA380 column in critically ill patients. | through study completion, an average of 24 months
  Number of patients unable to tolerate treatment with HA380 column.
Ability to recruit the sample size of eligible patients within the study period. | through study completion, an average of 24 months
  Proportion of the sample size recruited into the study during the study period.

SECONDARY OUTCOMES:
Time spent on vasopressor therapy. | From date admission to ICU, assessed up to 4 weeks
  Hours spent requiring vasopressor support.
Time spent in ICU | From date of admission to ICU until the date of ICU discharge or date of death, which ever comes first, assessed up to 24 months
  Days spent in ICU
ICU Mortality | From the date of admission to ICU until the date of death from any cause during ICU stay, assessed up to 24 months
  Death in ICU
Time spent on extracorporeal support | From the date of admission to ICU, assessed up to 24 weeks
  Days spent on extracorporeal support.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Granowitz EV, Clark BD, Mancilla J, Dinarello CA. Interleukin-1 receptor antagonist competitively inhibits the binding of interleukin-1 to the type II interleukin-1 receptor. J Biol Chem. 1991 Aug 5;266(22):14147-50. PMID 1830582
- [Background] Fisher CJ Jr, Dhainaut JF, Opal SM, Pribble JP, Balk RA, Slotman GJ, Iberti TJ, Rackow EC, Shapiro MJ, Greenman RL, et al. Recombinant human interleukin 1 receptor antagonist in the treatment of patients with sepsis syndrome. Results from a randomized, double-blind, placebo-controlled trial. Phase III rhIL-1ra Sepsis Syndrome Study Group. JAMA. 1994 Jun 15;271(23):1836-43. PMID 8196140
- [Background] Opal SM, Fisher CJ Jr, Dhainaut JF, Vincent JL, Brase R, Lowry SF, Sadoff JC, Slotman GJ, Levy H, Balk RA, Shelly MP, Pribble JP, LaBrecque JF, Lookabaugh J, Donovan H, Dubin H, Baughman R, Norman J, DeMaria E, Matzel K, Abraham E, Seneff M. Confirmatory interleukin-1 receptor antagonist trial in severe sepsis: a phase III, randomized, double-blind, placebo-controlled, multicenter trial. The Interleukin-1 Receptor Antagonist Sepsis Investigator Group. Crit Care Med. 1997 Jul;25(7):1115-24. doi: 10.1097/00003246-199707000-00010. PMID 9233735
- [Background] REMAP-CAP Investigators; Gordon AC, Mouncey PR, Al-Beidh F, Rowan KM, Nichol AD, Arabi YM, Annane D, Beane A, van Bentum-Puijk W, Berry LR, Bhimani Z, Bonten MJM, Bradbury CA, Brunkhorst FM, Buzgau A, Cheng AC, Detry MA, Duffy EJ, Estcourt LJ, Fitzgerald M, Goossens H, Haniffa R, Higgins AM, Hills TE, Horvat CM, Lamontagne F, Lawler PR, Leavis HL, Linstrum KM, Litton E, Lorenzi E, Marshall JC, Mayr FB, McAuley DF, McGlothlin A, McGuinness SP, McVerry BJ, Montgomery SK, Morpeth SC, Murthy S, Orr K, Parke RL, Parker JC, Patanwala AE, Pettila V, Rademaker E, Santos MS, Saunders CT, Seymour CW, Shankar-Hari M, Sligl WI, Turgeon AF, Turner AM, van de Veerdonk FL, Zarychanski R, Green C, Lewis RJ, Angus DC, McArthur CJ, Berry S, Webb SA, Derde LPG. Interleukin-6 Receptor Antagonists in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Apr 22;384(16):1491-1502. doi: 10.1056/NEJMoa2100433. Epub 2021 Feb 25. PMID 33631065
- [Background] Huang Z, Wang SR, Su W, Liu JY. Removal of humoral mediators and the effect on the survival of septic patients by hemoperfusion with neutral microporous resin column. Ther Apher Dial. 2010 Dec;14(6):596-602. doi: 10.1111/j.1744-9987.2010.00825.x. PMID 21118369
- [Background] Huang Z, Wang SR, Yang ZL, Liu JY. Effect on extrapulmonary sepsis-induced acute lung injury by hemoperfusion with neutral microporous resin column. Ther Apher Dial. 2013 Aug;17(4):454-61. doi: 10.1111/j.1744-9987.2012.01083.x. Epub 2012 Jun 21. PMID 23931889